CLINICAL TRIAL: NCT00291629
Title: Myocardial Regeneration and Angiogenesis in Myocardial Infarction With G-CSF and Intra-Coronary Stem Cell Infusion-3-DES (MAGIC Cell-3-DES)
Brief Title: Myocardial Regeneration and Angiogenesis in Myocardial Infarction With G-CSF and Intra-Coronary Stem Cell Infusion-3-DES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SeoulNUH cardiology
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; revascularization; drug eluting stents
MeSH Terms: conditions — Myocardial Infarction | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: G-CSF (Dong-A pharmaceutical, Seoul, Korea)
Procedure: collection of mobilized peripheral blood stem cells
Procedure: Intracoronary infusion of mobilized cells

SUMMARY:
This trial was performed to evaluate the safety of G-CSF based stem cell therapy and to compare outcome of intracoronary infusion of mobilized PBSCs between patients with AMI and OMI.

DETAILED DESCRIPTION:
The MAGIC Cell-DES trial was designed as a randomized, controlled trial to recruit 100 patients with AMI and OMI. Patients who were successfully revascularized with DES in the culprit lesion were eligible for enrollment. After revascularization, patients were randomized by use of a randomization table. After randomization, study processes were not blinded.

In the cell infusion groups after successful PCI, PBSCs were mobilized by daily subcutaneous injections of G-CSF (Dong-A pharmaceutical, Seoul, Korea) at 10 g/kg body weight for three days. At day 4, mobilized PBSCs were collected with COBE spectra apheresis system (COBE BCT. Inc., Lakewood, CO, USA) using the mononuclear cell collection methods and infused selectively to infarcted myocardium via over-the-wire balloon catheter.

The primary end point to evaluate efficacy was the change in LVEF, measured by MRI. The secondary end points were changes in LV volume, myocardial perfusion measured by coronary flow reserve (CFR), and the development of major adverse cardiac events (MACE; death, new MI, revascularization, hospitalization due to aggravation of ischemia or heart failure).

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute or old myocardial infarction who were successfully revascularized with DES in the culprit lesion were eligible for enrollment.

Exclusion Criteria:

* 1) Persistent severe heart failure (left ventricular ejection fraction (LVEF) < 20%) 2) Uncontrolled myocardial ischemia or ventricular tachycardia 3) Culprit lesion of infarct related artery not feasible for percutaneous coronary intervention (PCI) or unsuccessful PCI 4) Age > 80 years 5) Malignancy 6) Serious current infection or hematologic disease; and 7) Life expectancy under one year.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
the change in left ventricular ejection fraction (LVEF), which was measured by cardiac MRI | 6 month

SECONDARY OUTCOMES:
changes in left ventricular volume measured by echocardiography and MRI, myocardial perfusion by coronary flow reserve, and the development of major adverse cardiac events | 6month

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, Principal Investigator — Associated Professor of Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Yon-Gon Dong, Chongno-Gu, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Kang HJ, Kim HS, Zhang SY, Park KW, Cho HJ, Koo BK, Kim YJ, Soo Lee D, Sohn DW, Han KS, Oh BH, Lee MM, Park YB. Effects of intracoronary infusion of peripheral blood stem-cells mobilised with granulocyte-colony stimulating factor on left ventricular systolic function and restenosis after coronary stenting in myocardial infarction: the MAGIC cell randomised clinical trial. Lancet. 2004 Mar 6;363(9411):751-6. doi: 10.1016/S0140-6736(04)15689-4. PMID 15016484